CLINICAL TRIAL: NCT05403671
Title: Fit for Everyday Life - Increasing Exercise and Physical Activity in Those Rehablilitating From Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Lounais-Suomen Syöpäyhdistys (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: T0000/2022
Record Dates: First submitted 2022-05-10; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Cancer Survivor
Keywords: exercise; cancer survivor; rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Increasing Exercise and Physical Activity in Those Rehablilitating From Cancer — Intervention includes exercising and relaxation in a group

SUMMARY:
The aim of the study is to increase the physical activity and exercise of those recovering from cancer (after treatments) and to promote a functional return to everyday life and coping in everyday life. The aim of the study is to evaluate the effects of a exercise intervention on the quality of life, functional fitness (functional muscle strength and endurance tests) and the amount of physical activity of the participants in the study.

DETAILED DESCRIPTION:
Design: This is a quantitative study, whose data includes structured surveys (questionnaires) and measurements. Data are collected before and after the group exercise intervention. This 8 week tailored, progressive program will consist muscle strength training, endurance training, flexibility training, relaxation and home-exercises.

ELIGIBILITY:
Inclusion Criteria:

* Active cancer treatments have ended under 12 months
* Age 18-70 years
* Finnish speaking
* moving without aids
* z=1-0
* able to come Meri-Karina
* normal or low physical activity
* able to use digital equipments to participate remote exercise sessions

Exclusion Criteria:

* Exercise contraindications
* Memory and mental health problems
* Exercise every day over two hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The change of Quality of life | change from baseline at 8 weeks
  Eortec Qlqc-30
The change of Functional muscle strength | change from baseline at 8 weeks
  upper and lower body functionals muscle strength tests
The change of Endurance | change from baseline at 8 weeks
  6 min walking test
The change of Subjective physical activity | change from baseline at 8 weeks
  exercise diary
The change of Subjective physical capability | change from baseline at 8 weeks
  PROMIS-Cancer

SECONDARY OUTCOMES:
Experiences and feedback | only at 8 weeks
  subjective feedback survey

CONTACTS AND LOCATIONS:
Overall Officials: Pia Vihinen, MD, PhD, Study Director — Turku University Hospital
Locations (1):
- Maijastiina Rekunen, Turku, Finland

IPD SHARING:
Plan to Share IPD: No